CLINICAL TRIAL: NCT00226486
Title: Examination and Treatment of Elderly After a Fall- an Analysis in a Medical Technology Evaluation Perspective
Brief Title: Examination and Treatment of Elderly After a Fall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KA05059
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Accidental Falls

ARMS (2):
- 1 (Experimental): Identification of individual risk factors for falls and specified intervention aimed diminishing these risk factors in the individual.
  Interventions: Other: multifactorial intervention
- 2 (Placebo Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: multifactorial intervention — Identification of medical, cardiovascular, physical risk factors for falls; e.g. vision, drug-use, depression, carotid sinus syndrome, orthostatic hypotension, etc. Individual intervention; treatment of disease, drug review, pacemaker, exercises, new glasses, all if indicated.
  Arms: 1
Other: Usual care — No intervention, but ususal care after an accidental fall.
  Arms: 2

SUMMARY:
Falls and injurious falls are common among elderly people. The aim of the study is to test a model of multifactorial fall intervention in a Danish population of elderly sustaining a fall. Focus is on prevention of further falls, patients views on fall prevention and a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* Having been treated in emergency department or submitted to hospital after a fall
* Living in the Glostrup area.

Exclusion Criteria:

* Fall due to strong external force, new apoplexia cerebri, epileptic seizure, alcohol intoxication.
* Known cognitive impairment
* Not able to walk prior to fall
* Living in institution
* Planned geriatric intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 392 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Number of falls and injurious falls in 12 months

SECONDARY OUTCOMES:
Health related Quality of Life
Fear of falling
Dependence
Use of hospital, primary care etc.
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ane B Vind, Dr., Principal Investigator — Glostrup University Hospital
Locations (1):
- Department of Geriatrics, Amtssygehuset i Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Vind AB, Andersen HE, Pedersen KD, Joergensen T, Schwarz P. Effect of a program of multifactorial fall prevention on health-related quality of life, functional ability, fear of falling and psychological well-being. A randomized controlled trial. Aging Clin Exp Res. 2010 Jun;22(3):249-54. doi: 10.1007/BF03324804. Epub 2009 Nov 17. PMID 19934621